CLINICAL TRIAL: NCT05681221
Title: Clinical and Radiographic Evaluation of the Synergistic Effect of Nano Silver Particles and Calcium Hydroxide Versus Triple Antibiotic Paste as Antibacterial Agents for Lesion Sterilization and Tissue Repair (LSTR) in Necrotic Primary Molars: Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of the Synergistic Effect of Nano Silver Particles and Calcium Hydroxide Versus Triple Antibiotic Paste as Antibacterial Agents for Lesion Sterilization and Tissue Repair (LSTR) in Necrotic Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sohair Magdy Abdel Fattah Aly, Pediatric Resident at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSTR
Record Dates: First submitted 2022-12-13; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Root Canal Infection
Keywords: primary teeth; LSTR; necrotic
MeSH Terms: conditions — Necrosis | interventions — Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: TAP is an efficient antibacterial for the disinfection of the periapical area in the necrotic primary second molars as well as the infected dentinal tubules. It is effective against the persistent odontogenic infections.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSTR in necrotic primary second molar using TAP (Active Comparator): Triple antibiotic paste (TAP) is considered the gold standard in LSTR. It is a combination of ciprofloxacin, metronidazole and minocycline. Many anaerobic bacteria are resistant to ciprofloxacin. Hence, it is often used with metronidazole in treating mixed infections to compensate for its limited scope. Therefore, TAP can affect gram-negative, gram-positive, and anaerobic bacteria, and this combination can be effective against odontogenic microorganisms.
  Interventions: Other: TAP
- LSTR in necrotic primary second molar using nano silver particles and calcium hydroxide (Experimental): Nano silver particles have a strong anti-bacterial properties due to its ability to target the bacteria on different cellular levels. Calcium hydroxide has been used for so long as an intra canal medication in odontogenic infections due to its strong alkalinity that gives it its anti bacterial properties. This combination might be a future alternative to antibiotics, in an attempt to decrease the bacterial antibiotic resistance and antibiotics use.
  Interventions: Other: Nano silver particles and calcium hydroxide

INTERVENTIONS:
Other: Nano silver particles and calcium hydroxide — Combination of two materials that can possibly eradicate the mixed odontogenic infection in the periapical area and dentinal tubules in necrotic primary second molars.
  Arms: LSTR in necrotic primary second molar using nano silver particles and calcium hydroxide
Other: TAP — Triple antibiotic paste (TAP) is considered the gold standard in LSTR. It is a combination of ciprofloxacin, metronidazole and minocycline. Many anaerobic bacteria are resistant to ciprofloxacin. Hence, it is often used with metronidazole in treating mixed infections to compensate for its limited scope. Therefore, TAP can affect gram-negative, gram-positive, and anaerobic bacteria, and this combination can be effective against odontogenic microorganisms.
  Arms: LSTR in necrotic primary second molar using TAP

SUMMARY:
Could the clinical and radiographic success of Nano Silver Particles and Calcium Hydroxide be comparable to that of Triple Antibiotic Paste as antibacterial agents for Lesion Sterilization and Tissue Repair (LSTR) in necrotic second primary molars?

DETAILED DESCRIPTION:
The major aim of pediatric dentistry is to maintain the integrity of the primary dentition until physiologic exfoliation. Premature loss of primary teeth may lead to several complications, like disturbance in eruption sequence, ectopic eruption and space loss. Hence, the conservation of primary tooth structure is essential, provided that it can be restored to function and remain free from disease.Pulp therapy in primary teeth at times become contraindicated or compromised due to excessive root resorption, inadequate bone and periodontal support, a child with pre-cooperative age group, etc.

In the current era, a new perspective which is less invasive and less time consuming procedure could be a spark of hope for pedodontists. The Lesion Sterilization and Tissue Repair (LSTR) claims its significance in such clinical situation. The concept of LSTR was developed at the Cariology Research Unit of Niigata University School of Dentistry. The LSTR is an endodontic treatment procedure that involves non instrumentation or minimal instrumentation followed by placement of antibiotic mixture to disinfect root canal systems, and periapical lesions. The basic concept of LSTR is "do not remove or touch and leave it.". The principle behind LSTR is repair by natural defense mechanisms of host; Sterilizing the root canals and pulp chamber by medicaments can decrease the bacterial load. If the procedure is successful tissue repair can be expected.

However, because it is impossible to eradicate all microorganisms from the root canal system throughout the treatment, endodontic materials must contain specific components that release antibacterial substances. The most likely cause for this is the complex anatomy of the root canal system, which allows bacteria to colonize in inaccessible places to antimicrobial agents. Despite cleaning, and administration of highly effective antimicrobial agents, clinical trials have shown that bacteria remain within the root canal system because bacteria can form biofilms, infiltrate dentinal tubules, and cause monoinfection.

Among the intra canal medicaments, calcium hydroxide is most frequently used because of its wide antimicrobial spectrum. Calcium hydroxide Ca(OH)2 is commonly employed as an intra canal medicament. It releases hydroxyl ions which causes high alkalinity. Nevertheless, the ability of calcium hydroxide in elimination of bacteria from the root canal has been questioned. Antibacterial ability of calcium hydroxide in aqueous environment is linked to the discharge of hydroxyl ions. It can cause damage to the cytoplasmic membrane, bacterial DNA as well as can cause protein denaturation.

However, calcium hydroxide is not as much effective when used for canal disinfection having established Enterococcus faecalis (E.faecalis) biofilm. Recently, numerous studies have introduced silver nanoparticles as an antimicrobial agent. Silver nanoparticles have antimicrobial activity and are biocompatible, silver ions can cause damage to the bacterial cell wall. These are productive against many microorganisms including E.faecalis. Nanoparticles have /polyanionic polycationic properties with a high surface area and positive charge density, which increases their antibacterial activity. The particle size was also related to antimicrobial activity; the smaller particles give more bactericidal effects compared to larger particles. Calcium hydroxide do not always eradicate E.faecalis biofilm from root canals. Hence, it is essential to introduce advanced endodontic intra-canal medicament approaches that are successful in eradicating biofilm bacteria inside the root canals.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 years and 7 years.
* Restorable necrotic mandibular second primary molars
* Mandibular lower second primary molar with signs of radiolucency in periapical or furcation area.
* Mandibular lower second primary molar with widening of PDL space or loss of lamina dura continuity.
* Mandibular lower second primary molar with evidence of internal/external pathologic root resorption.

Signs of radiolucency in periapical or furcation area.

* Widening of PDL space or loss of lamina dura continuity.
* Evidence of internal/external pathologic root resorption.
* External root resorption from 1% to 50%.

Exclusion Criteria:

* Children that are not apparently healthy.
* Lack of informed consent by the child patient's parent.
* Patients allergic to any antibiotic used in the preparation of the TAP.
* Unable to attend follow-up visits.
* Refusal of participation.
* External root resorption above 50%.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological mobility | 1 year.
  presence/ absence. Mobility test by applying pressure using the handle of dental mirrors
Post-operative pain | 1 year.
  presence/ absence. Verbal question to patient/ parent.
Soft tissue pathology | 1 year.
  presence/ absence. Visual clinical examination
Pain to percussion | 1 year.
  presence/ absence. Percussion test by the handle of the dental mirror

SECONDARY OUTCOMES:
Absence of furcation or periapical radiolucency | 1 year.
  Intra-oral digital peri-apical x-ray
Absence of external or internal root resorption | 1 year.
  Intra-oral digital peri-apical x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Rania A. Nasr, PhD, Study Chair — Cairo University

REFERENCES:
- [Background] Shetty A, Geethanjali G, Hegde A. Lesion sterilization and tissue repair in primary teeth. SRM Journal of Research in Dental Sciences. 2020;11(2):99. doi:10.4103/srmjrds.srmjrds_87_19
- [Background] Takushige T, Cruz EV, Asgor Moral A, Hoshino E. Endodontic treatment of primary teeth using a combination of antibacterial drugs. Int Endod J. 2004 Feb;37(2):132-8. doi: 10.1111/j.0143-2885.2004.00771.x. PMID 14871180
- [Background] Motiwala MA, Habib S, Ghafoor R, Irfan S. Comparison of antimicrobial efficacy of Calcipex and Metapex in endodontic treatment of chronic apical periodontitis: a randomised controlled trial study protocol. BMJ Open. 2021 Jul 21;11(7):e048947. doi: 10.1136/bmjopen-2021-048947. PMID 34290069
- [Background] Mohammadi Z, Shalavi S, Yazdizadeh M. Antimicrobial activity of calcium hydroxide in endodontics: a review. Chonnam Med J. 2012 Dec;48(3):133-40. doi: 10.4068/cmj.2012.48.3.133. Epub 2012 Dec 21. PMID 23323217
- [Background] Afkhami F, Pourhashemi SJ, Sadegh M, Salehi Y, Fard MJ. Antibiofilm efficacy of silver nanoparticles as a vehicle for calcium hydroxide medicament against Enterococcus faecalis. J Dent. 2015 Dec;43(12):1573-9. doi: 10.1016/j.jdent.2015.08.012. Epub 2015 Aug 29. PMID 26327612
- [Background] Zapór L. Effects of silver nanoparticles of different sizes on cytotoxicity and oxygen metabolism disorders in both reproductive and respiratory system cells. Archives of Environmental Protection. 2016;42(4):32-47. doi:10.1515/aep-2016-0038
- [Background] Riaz Z, Raza M, Hanif A, Haider B, Akram S, Safdar S. Antibacterial efficacy of silver nanoparticles impregnated calcium hydroxide: An in vitro study. J Pak Dent Assoc 2022;31(1):1-4
- [Background] Deepak BM, Prabhakar AR, Karuna YM, Sugandhan S, Zahoor N, Mahendrapa Shagale A. Evaluation of the Antibacterial Activity of Triclosan-incorporated Root Canal Filling Materials for Primary Teeth against Enterococcus faecalis. Int J Clin Pediatr Dent. 2021 May-Jun;14(3):393-397. doi: 10.5005/jp-journals-10005-1960. PMID 34720513